CLINICAL TRIAL: NCT01445626
Title: A Retrospective Data Collection Study in Patients Receiving Dexamethasone Intravitreal Implant (Ozurdex®) for Macular Oedema Due to Retinal Vein Occlusion (RVO)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/RET/010
Record Dates: First submitted 2011-09-30; First posted 2011-10-04 (Estimated); Results first posted 2013-02-18 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-01

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: Patients who received at least two OZURDEX® (dexamethasone intravitreal implant) injections.
  Interventions: Drug: dexamethasone intravitreal implant 0.7 mg

INTERVENTIONS:
Drug: dexamethasone intravitreal implant 0.7 mg — Dexamethasone intravitreal implant 0.7 mg was dosed previously according to general clinical practice.
  Other Names: OZURDEX®

SUMMARY:
This study will use retrospective data to evaluate the efficacy, safety, and re-injection interval of OZURDEX® in the treatment of macular oedema due to Retinal Vein Occlusion (RVO).

ELIGIBILITY:
Inclusion Criteria:

* Macular oedema in the study eye due to BRVO or CRVO
* Received at least 2 OZURDEX® injections in the study eye

Exclusion Criteria:

* Received OZURDEX® injections as part of or during any clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received at least 2 injections of OZURDEX® to treat macular oedema due to branch retinal vein occlusion (BRVO) or central retinal vein occlusion (CRVO) in at least 1 eye.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Münster, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 87
Completed | 87
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 87
Age Continuous [Mean (Standard Deviation); unit: Years] — Age Mean and Standard Deviation is based on data available for 83 patients. Age data is missing for 4 patients.
  Years | 68.48 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 58

OUTCOME MEASURES:

1. Primary Outcome: Time to OZURDEX® Re-injection
Description: Time to OZURDEX® re-injection is the time in days between the first and second OZURDEX® injections.
Time Frame: Up to 12 months
Population: All participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | All Participants
Number analyzed (Participants) | 85
Days | 140.80 (56.65) [28.0 to 323.0]

2. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) 7 to 12 Weeks Following the Last Injection
Description: BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of letters ranging from 0 (worse) to 100 (best). The change in BCVA was calculated using the most improved number of letters read correctly between 7 and 12 weeks following the last injection of OZURDEX® - the number of letters read correctly at baseline. A positive change from baseline indicates improvement.
Time Frame: Baseline, 7 to 12 weeks following the last injection
Population: All participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | All Participants
Number analyzed (Participants) | 35
Letters
  Baseline | 50.97 (18.82) [20.0 to 76.0]
  Change from baseline 7-12 wks after last injection | 10.89 (21.21) [-41.0 to 45.0]

3. Secondary Outcome: Percentage of Patients With an Increase of 2 Lines or More in BCVA
Description: BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worse) to 20 (best). An increase of 2 or more lines read correctly compared to baseline is an improvement.
Time Frame: Baseline, Up to 12 months
Population: All treated participants.
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 87
Percentage of participants | 56.3

4. Secondary Outcome: Percentage of Patients With an Increase of 3 Lines or More in BCVA
Description: BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worse) to 20 (best). An increase of 3 or more lines read correctly compared to baseline is an improvement.
Time Frame: Baseline, Up to 12 months
Population: All treated participants.
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 87
Percentage of participants | 50.6

5. Secondary Outcome: Change From Baseline in Central Retinal Thickness by Optical Coherence Tomography (OCT) 7 to 12 Weeks Following the Last Injection
Description: Optical Coherence Tomography (OCT), a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina, was performed in the study eye after pupil dilation at baseline and 7 to 12 weeks after the last injection. A negative change from baseline indicates improvement.
Time Frame: Baseline, 7 to 12 weeks following the last injection
Population: All participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | All Participants
Number analyzed (Participants) | 34
µm
  Baseline | 576.85 (204.66)
  Change from baseline 7-12 wks after last injection | -259.21 (265.35)

6. Secondary Outcome: Time to Improvement of 2 Lines or More in BCVA
Description: Time to improvement of 2 lines or more in BCVA is defined as the number of days after the first injection of OZURDEX® to achieve an improvement of 2 or more lines read correctly compared to baseline. BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worse) to 20 (best).
Time Frame: Baseline, Up to 12 months
Population: All participants with data available for analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | All Participants
Number analyzed (Participants) | 42
Days | 55.0 [27.0 to 184.0]

7. Secondary Outcome: Time to Improvement of 3 Lines or More in BCVA
Description: Time to improvement of 3 lines or more in BCVA is defined as the number of days after the first injection of OZURDEX® to achieve an improvement of 3 or more lines read correctly compared to baseline. BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worse) to 20 (best).
Time Frame: Baseline, Up to 12 months
Population: All participants with data available for analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | All Participants
Number analyzed (Participants) | 35
Days | 57.0 [27.0 to 208.0]

ADVERSE EVENTS:
Description: This was a retrospective study. Patient charts were reviewed for adverse events (AEs). All AEs related to study drug were collected from the time of the first OZURDEX® injection through six months after the last injection.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 6/87
Other Adverse Events (participants affected / at risk) | 47/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=87)
Cataract operation (Eye disorders) | 3
Suspected glaucoma (Eye disorders) | 1
Choroidal detachment (Eye disorders) | 1
Cataract progression (Eye disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=87)
Intraocular pressure increased (Investigations) | 16
Glaucoma (Eye disorders) | 10
Eye laser surgery (Eye disorders) | 9
Cataract operation (Eye disorders) | 6
Retinal degeneration (Eye disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.